CLINICAL TRIAL: NCT04804631
Title: A Mixed Methods Study Investigating Complications, Outcomes and Family Experiences of Gastrostomy Feeding in Paediatric Allogeneic Bone Marrow Transplantation
Brief Title: Tube Feeding in Children Having a Bone Marrow Transplant
Status: Completed | Type: Observational
Sponsor: Institute of Child Health (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 19SH04
Record Dates: First submitted 2021-02-09; First posted 2021-03-18 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Bone Marrow Disease; Stem Cell Transplant Complications; Enteral Feeding Intolerance; Gastrostomy; Gastrostomy Complications; Experiences, Life
Keywords: Bone marrow transplantation; Haematopoietic stem cell transplantation; Nasogastric tube; Nutritional status
MeSH Terms: conditions — Bone Marrow Diseases | interventions — Enteral Nutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gastrostomy tube: Prophylactic gastrostomy placed prior to bone marrow transplant.
  Interventions: Device: Enteral feeding tubes
- Nasogastric tube: Nasogastric tube placed during admission.
  Interventions: Device: Enteral feeding tubes

INTERVENTIONS:
Device: Enteral feeding tubes — Families within Great Ormond Street Hospital are offered the choice of two enteral feeding tubes prior to admission for bone marrow transplant. Some families choose a gastrostomy to be placed prophylactically in the weeks prior to admission, others choose a nasogastric tube to be placed during the admission.

SUMMARY:
The purpose of this study is to assess the problems and a range of nutritional and clinical outcomes that occur with two feeding tubes used by children having a bone marrow transplant. Children and parents will also be interviewed to ask about their experiences of tube feeding.

DETAILED DESCRIPTION:
Background: Bone marrow transplant (BMT) is the only potentially curative treatment for children with malignant and non-malignant diseases. Chemotherapy provided during BMT causes side-effects including diarrhoea and vomiting meaning all children become unable to eat and require tube feeding. All 16 centres in the UK use a nasogastric tube. Great Ormond Street Hospital offer families a gastrostomy as an alternative. Minimal published literature exists on gastrostomies in this population.

Aims: Investigate complications, outcomes and family experiences of gastrostomy tubes in paediatric BMT.

Objectives:

1. Survey current nutrition practices, use and opinions towards gastrostomy tubes in UK paediatric BMT centres.
2. Compare clinical outcomes and complications occurring from gastrostomy versus nasogastric tubes in children during BMT.
3. Investigate decision making and experiences of families regarding tube feeding.

Methods: A multiphase, convergent parallel mixed methods study across 3 work packages (WPs).

1. Survey: A survey will be sent to a dietitian, nurse and doctor (the staff involved in tube feeding) in each UK paediatric BMT centre. Questions will focus on nutrition practices, and current use and opinions of gastrostomies.
2. Prospective cohort study: Outcomes will be compared between children fed via gastrostomy versus nasogastric tube from admission to six months post-BMT. All children transplanted over one year at one centre will be included. Outcomes including complications occurring with both tubes, dietary intake and anthropometry will be investigated. Anticipated sample size is 9-15 children fed via gastrostomy, 30-50 via nasogastric tube.
3. Family interviews: Families from WP 2 will be invited to be interviewed at two times; on admission to discuss why they did or did not choose a gastrostomy, and one month after discharge to discuss their experience of tube feeding. Creative methods including drawing and scrapbooks will be used during children's interviews to help them articulate their thoughts. Parents will take part in semi-structured interviews.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the centre during the study period for an allogeneic bone marrow transplant (BMT) for any diagnosis.
* Receiving any conditioning regimen, donor type and stem cell source.
* Children admitted for their second or more BMT.
* Children admitted on an established enteral tube feeding regimen.
* NHS patients.

Exclusion Criteria:

* Children receiving first-line, prophylactic, parenteral nutrition as this is not the standard nutrition pathway of most children receiving BMT at the centre. This is usually given in specific circumstances such as children receiving cord blood transplants or those with gastrointestinal diseases.
* Autologous BMT, including children receiving chimeric antigen receptor T-cell therapy (CAR-T).
* No feeding tube placed and no nutrition support required from tube feeding or parenteral nutrition. Children rarely do not require any form of nutrition support.

Ages: 1 Month to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children admitted to the centre over 12 months (allowing six months follow up) for an allogeneic BMT, for any diagnosis (malignant or non-malignant), planned to receive any type of conditioning and any donor type, will be eligible and vetted according to the inclusion/exclusion criteria. Children transplanted at the centre mainly come from London, but can be from other parts of the UK too, and are anywhere between a few months old up to the eldest of around 13 years.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Weight Z-score | Measured weekly for six weeks from admission for bone marrow transplant, and monthly thereafter to six months post-transplant (6 months)
  Change in weight Z-score between groups. Measured using ward scales.

SECONDARY OUTCOMES:
Gastrostomy tube complications | Measured weekly for six weeks from admission for bone marrow transplant, and monthly thereafter to tube removal or six months post-transplant, whichever comes first (6 months)
  Categorical reporting of the incidence of any complications occurring with the gastrostomy tube e.g. infection, dislodgement, blockage
Nasogastric tube complications | Measured weekly for six weeks from admission for bone marrow transplant, and monthly thereafter to tube removal or six months post-transplant, whichever comes first (6 months)
  Categorical reporting of the incidence of any complications occurring with the nasogastric tube e.g. dislodgement, blockage
Height Z-score | Measured monthly from admission to six months post-transplant (6 months)
  Change in height Z-score between groups. Measured using ward stadiometer.
Body mass index (BMI) Z-score | Measured monthly from admission to six months post-transplant (6 months)
  Change in BMI Z-score between groups. Weight and height will be combined to report BMI in kg/m^2 and converted to Z-scores.
Mid-upper-arm circumference (MUAC) Z-score | Measured weekly for six weeks from admission for bone marrow transplant, and monthly thereafter to six months post-transplant (6 months)
  Change in MUAC Z-score between groups. Measured using ward measuring tape.
Overall survival | Measured for all children at day-100 post-transplant
  Percentage of children alive (with death from any cause) 100 days post-bone marrow transplant
Non-relapse mortality | Measured for all children at day-100 post-transplant
  Percentage of children alive (with death not caused by disease relapse) 100 days post-bone marrow transplant
Graft-versus-host disease grade III-IV | Measured for all children at day-100 post-transplant
  Percentage of children with grade III-IV graft-versus-host disease (measured using modified Gluckberg classification) 100 days post-bone marrow transplant
Gastrointestinal graft-versus-host disease | Measured for all children at day-100 post-transplant
  Percentage of children with gut graft-versus-host disease (measured using modified Gluckberg classification) 100 days post-bone marrow transplant
Calorie intake | Measured weekly for six weeks from admission for bone marrow transplant, and monthly thereafter to six months post-transplant (6 months)
  Average intake of calories (total kcal intake and kcals/kg) provided from oral, enteral and parenteral nutrition, averaged over 3-days, measured from the hospital's electronic patient records during the bone marrow transplant admission, and thereafter once the child is at home from 3-day food diaries recorded once per month.
Protein intake | Measured weekly for six weeks from admission for bone marrow transplant, and monthly thereafter to six months post-transplant (6 months)
  Average intake of protein (total protein intake and grams/kg) provided from oral, enteral and parenteral nutrition, averaged over 3-days, measured from the hospital's electronic patient records during the bone marrow transplant admission, and thereafter once the child is at home from 3-day food diaries recorded once per month.
Fluid intake | Measured weekly for six weeks from admission for bone marrow transplant, and monthly thereafter to six months post-transplant (6 months)
  Average intake of fluid (total fluid intake and ml/kg) provided from oral, enteral and parenteral nutrition, averaged over 3-days, measured from the hospital's electronic patient records during the bone marrow transplant admission, and thereafter once the child is at home from 3-day food diaries recorded once per month.
Duration of enteral nutrition | Measured from admission for bone marrow transplant to tube removal or discharge home post-transplant, whichever comes first. (Hospital admission is usually 3 months)
  Total number of days enteral nutrition is provided during admission for bone marrow transplant
Duration of parenteral nutrition | Measured from admission for bone marrow transplant to tube removal or discharge home post-transplant, whichever comes first. (Hospital admission is usually 3 months)
  Total number of days parenteral nutrition is provided during admission for bone marrow transplant
Use of enteral feeding tube | Measured weekly for six weeks from admission for bone marrow transplant, and monthly thereafter to six months post-transplant (6 months)
  Categorical description of what the enteral feeding tube is used for. Categories include: "Not in use", "Nutrition only", "Medicines only", "Fluids only", "Nutrition & medicines", "Medicines & fluids", "Nutrition, medicines & fluids".
Blood copper level | Measured monthly from admission for bone marrow transplant until the child is discharged home following the transplant (hospital admission is usually 3 months)
  Change in blood copper level (micromol/L) during admission for bone marrow transplant
Blood selenium level | Measured monthly from admission for bone marrow transplant until the child is discharged home following the transplant (hospital admission is usually 3 months)
  Change in blood selenium level (micromol/L) during admission for bone marrow transplant
Blood zinc level | Measured monthly from admission for bone marrow transplant until the child is discharged home following the transplant (hospital admission is usually 3 months)
  Change in blood zinc level (micromol/L) during admission for bone marrow transplant
Blood vitamin A level | Measured monthly from admission for bone marrow transplant until the child is discharged home following the transplant (hospital admission is usually 3 months)
  Change in blood vitamin A level (micromol/L) during admission for bone marrow transplant
Blood vitamin E level | Measured monthly from admission for bone marrow transplant until the child is discharged home following the transplant (hospital admission is usually 3 months)
  Change in blood vitamin E level (micromol/L) during admission for bone marrow transplant

CONTACTS AND LOCATIONS:
Overall Officials: Faith Gibson, Professor, Principal Investigator — Great Ormond Street Hospital
Locations (1):
- Great Ormond Street Hospital, London, United Kingdom

REFERENCES:
- [Background] Evans J, Needle JJ, Hirani SP. Early outcomes of gastrostomy feeding in paediatric allogenic bone marrow transplantation: A retrospective cohort study. Clin Nutr ESPEN. 2019 Jun;31:71-79. doi: 10.1016/j.clnesp.2019.02.014. Epub 2019 Mar 21. PMID 31060837
- [Background] Gonzales F, Bruno B, Alarcon Fuentes M, De Berranger E, Guimber D, Behal H, Gandemer V, Spiegel A, Sirvent A, Yakoub-Agha I, Nelken B, Duhamel A, Seguy D. Better early outcome with enteral rather than parenteral nutrition in children undergoing MAC allo-SCT. Clin Nutr. 2018 Dec;37(6 Pt A):2113-2121. doi: 10.1016/j.clnu.2017.10.005. Epub 2017 Oct 12. PMID 29097037
- [Background] Hoffmeister PA, Storer BE, Macris PC, Carpenter PA, Baker KS. Relationship of body mass index and arm anthropometry to outcomes after pediatric allogeneic hematopoietic cell transplantation for hematologic malignancies. Biol Blood Marrow Transplant. 2013 Jul;19(7):1081-6. doi: 10.1016/j.bbmt.2013.04.017. Epub 2013 Apr 25. PMID 23623893
- [Background] Trehan A, Viani K, da Cruz LB, Sagastizado SZ, Ladas EJ. The importance of enteral nutrition to prevent or treat undernutrition in children undergoing treatment for cancer. Pediatr Blood Cancer. 2020 Jun;67 Suppl 3:e28378. doi: 10.1002/pbc.28378. PMID 32614140
- [Background] McGrath KH, Hardikar W. Gastrostomy tube use in children with cancer. Pediatr Blood Cancer. 2019 Jul;66(7):e27702. doi: 10.1002/pbc.27702. Epub 2019 Mar 11. PMID 30854790
- [Background] Williams-Hooker R, Adams M, Havrilla DA, Leung W, Roach RR, Mosby TT. Caregiver and health care provider preferences of nutritional support in a hematopoietic stem cell transplant unit. Pediatr Blood Cancer. 2015 Aug;62(8):1473-6. doi: 10.1002/pbc.25473. Epub 2015 Mar 21. PMID 25809410
- [Background] Peric Z, Botti S, Stringer J, Krawczyk J, van der Werf S, van Biezen A, Aljurf M, Murray J, Liptrott S, Greenfield DM, Duarte RF, Ruutu T, Basak GW. Variability of nutritional practices in peritransplant period after allogeneic hematopoietic stem cell transplantation: a survey by the Complications and Quality of Life Working Party of the EBMT. Bone Marrow Transplant. 2018 Aug;53(8):1030-1037. doi: 10.1038/s41409-018-0137-1. Epub 2018 Mar 7. PMID 29515252